CLINICAL TRIAL: NCT02637232
Title: Mirvaso® Utilisation and Patient Satisfaction Evaluation
Brief Title: Mirvaso® Utilisation and Patient Satisfaction Evaluation (MUSE)
Acronym: MUSE
Status: Completed | Type: Observational
Sponsor: Galderma R&D (Industry)
Collaborators: Chiltern International Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RD.03.SPR.104160
Record Dates: First submitted 2015-12-16; First posted 2015-12-22 (Estimated); Results first posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea | interventions — Brimonidine Tartrate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mirvaso® / Onreltea TM
  Interventions: Other: Mirvaso® / Onreltea TM

INTERVENTIONS:
Other: Mirvaso® / Onreltea TM

SUMMARY:
The aim of the study is to evaluate the level of satisfaction among patients to whom Mirvaso® / Onreltea TM (trade mark) is prescribed.

ELIGIBILITY:
Inclusion Criteria:

* Patients to whom the physician has already decided to prescribe Mirvaso® /OnrelteaTM according to package insert

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with persistent facial erythema of rosacea
Sampling Method: Non-Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2015-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Investigator site 1, Hamilton, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Mirvaso® / Onreltea TM: Mirvaso® / Onreltea TM
Period: Overall Study
Arm/Group | Mirvaso® / Onreltea TM
Started | 301
Completed | 246
Not Completed | 55
Not completed — Lost to Follow-up | 42
Not completed — Adverse Event | 11
Not completed — patient 's decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Mirvaso® / Onreltea TM
Number analyzed (Participants) | 301
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.4 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 218
  Male | 83
Duration of rosacea [Mean (Standard Deviation); unit: Years] | 5.5 (7.9)
Previous therapies in the last 2 years [Count of Participants; unit: Participants] | 150
Subject previously prescribed by Mirvaso [Count of Participants; unit: Participants] | 65
Severity of facial erythema (by physician) [Count of Participants; unit: Participants]
  Mild | 68
  Moderate | 179
  Severe | 53
  Missing | 1
Severity of facial erythema (by subject) [Count of Participants; unit: Participants]
  Mild | 58
  Moderate | 169
  Severe | 73
  Missing | 1
Additional signs and Symptoms [Count of Participants; unit: Participants] — Population: Each subject can present several signs and symptoms. Here, number analyzed=participants with available data for specified categories.
  Participants
    Flushing present: number analyzed (Participants) | 298
    Flushing present | 250
    Papules and Pustules: number analyzed (Participants) | 298
    Papules and Pustules | 127
    Skin burning & stinging sensation: number analyzed (Participants) | 298
    Skin burning & stinging sensation | 151
    Rhinophyma: number analyzed (Participants) | 298
    Rhinophyma | 16
    Ocular manifestation: number analyzed (Participants) | 298
    Ocular manifestation | 29
    Telangiectasis: number analyzed (Participants) | 298
    Telangiectasis | 205
    Other signs and symptoms: number analyzed (Participants) | 298
    Other signs and symptoms | 1

OUTCOME MEASURES:

1. Primary Outcome: Satisfaction Among Patients to Whom Mirvaso®/OnrelteaTM is Prescribed Question
Time Frame: Week 4
Population: Analysis was performed on total population. Here, "Overall Number of Participants Analyzed" = participants with available data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Mirvaso® / Onreltea TM
Number analyzed (Participants) | 237
Participants
  Very satisfied | 55
  Somewhat satisfied | 86
  Neither satisfied nor dissatisfied | 38
  Somewhat dissatisfied | 31
  Very dissatisfied | 27

ADVERSE EVENTS:
Time Frame: From Baseline (Day 0) up to study follow-up visit at Week 4 (Day 31).
Description: Analysis was performed on safety population that comprised of subjects included and with at least a post-Baseline visit or information regarding the adverse event.
Arm/Group | Mirvaso® / Onreltea TM
All-Cause Mortality (participants affected / at risk) | 0/259
Serious Adverse Events (participants affected / at risk) | 1/259
Other Adverse Events (participants affected / at risk) | 61/259
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirvaso® / Onreltea TM (N=259)
ANGINA PECTORIS (Cardiac disorders) | 1 (1)
AORTIC ECTASIA (Vascular disorders) | 1 (1)
STENOSIS OF ILIACA EXTERNAL (Vascular disorders) | 1 (1)
RIVA STENOSIS (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirvaso® / Onreltea TM (N=259)
Erythema (Skin and subcutaneous tissue disorders) | 32 (36)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (7)
Rosacea (Skin and subcutaneous tissue disorders) | 8 (8)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 33 (36)
Skin irritation (Skin and subcutaneous tissue disorders) | 17 (17)
Flushing (Vascular disorders) | 30 (30)
Skin swelling (Skin and subcutaneous tissue disorders) | 7 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This is an agreement between the PI and sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed. Disclosure agreement is covered by a contract.